CLINICAL TRIAL: NCT07325253
Title: A Pilot Study to Correlate 4-18F- Fluoro-1-naphthol 18F-4FN PET/CT Imaging With Chronic Graft Versus Host Disease Manifestations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-1051; NCI-2026-00037 (Other: NCI-CTRP Clinical Registr)
Record Dates: First submitted 2026-01-06; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Pilot Study; PET/CT Imaging; Host Disease Manifestation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 (Experimental): Prognostic Biomarker Analysis - [18F]4FN PET/CT at Baseline
  Interventions: Drug: [18F]-4FN; Other: PET-CT
- Part 2 (Experimental): Predictive/PD Biomarker Analysis - [18F]4FN PET/CT before a New Systemic Therapy
  Interventions: Drug: [18F]-4FN; Other: PET-CT

INTERVENTIONS:
Drug: [18F]-4FN — Given by IV
Other: PET-CT — Imaging

SUMMARY:
To study the safety and possible side effects of using the imaging agent 4-[18F]Fluoro-1-Naphthol (also called [18F]4FN) in PET/CT scans for participants with chronic GVHD.

DETAILED DESCRIPTION:
Primary Objective

Determine the spatial and temporal correlation between [18F]4FN PET/CT measurements and the clinical manifestations and severity of chronic GVHD. We hypothesize that [18F]4FN PET/CT imaging features will anatomically and by intensity (SUV) correlate with concurrent chronic GVHD manifestations. We also hypothesize that PET/CT imaging features will temporally precede chronic GVHD manifestations at target anatomic locations.

ELIGIBILITY:
Eligibility Criteria

1. Chronic GVHD involving the joints, defined as any limitation of range of motion measured by Photographic Range Of Motion (PROM). Criteria can be found at (Jagasia, et al. 2015).
2. Able to give written informed consent.
3. ≥18 years of age
4. Creatinine clearance ≥ 30 mL/min/1.73m2
5. Non-joint chronic GVHD diagnostic / distinctive features are allowed.
6. Subjects may be planned to receive a new systemic therapy for chronic GVHD
7. Prior/continuing systemic therapy for chronic GVHD is allowed
8. ECOG performance status ≤2
9. Ability to understand and the willingness to sign a written informed consent document.
10. The effects of the study agent on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following:

    * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
    * History of hysterectomy or bilateral salpingo-oophorectomy.
    * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
    * History of bilateral tubal ligation or another surgical sterilization procedure.

      * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
11. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study agent administration.

Exclusion Criteria

1. Unable to comply with all study procedures (for example, participants who are unable to come to all follow up visits because they live far away from the transplant center)
2. Pregnant or lactating women: pregnant women are excluded from this study because the effects of [18F]4FN in pregnancy are not known.
3. Subjects with contraindications to the use of [18F]4FN including confirmed allergy.
4. Participants with a body weight of 400 pounds or more, or a body habitus which precludes their entry into the bore of the PET/CT scanner, because the hardware is not intended to support that weight.
5. Any additional medical condition, serious concurrent illness, or other extenuating circumstance that, in the opinion of the investigator, may significantly interfere with study compliance.
6. Children below the age of 18 are excluded because of the unknown but potential risks of administration of radiopharmaceuticals to minors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2028-01-03 (Estimated); Study Completion 2030-01-03 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs). | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: George L Chen, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org